CLINICAL TRIAL: NCT04428112
Title: Evaluating the Effectiveness of an Online Small-Group Self-Management Workshop for Rural Caregivers of Individuals With Alzheimer's Disease and Related Dementias
Brief Title: Rural Dementia Caregiver Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18-25814; 5R01AG057855-02 (NIH); 3R01AG057855-02S1 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Depression; Stress, Psychological; Self Efficacy; Loneliness; Social Isolation; Health Care Utilization; Dementia; Dementia Alzheimers; Dementia of Alzheimer Type; Dementia, Vascular; Dementia Frontal; Dementia, Lewy Body; Dementia, Mixed; Dementia in Parkinsons Disease; Dementia, HIV; Dementia Frontotemporal; Dementia, Multi-Infarct
Keywords: Caregiver; Caregiving
MeSH Terms: conditions — Depression; Stress, Psychological; Social Isolation; Patient Acceptance of Health Care; Dementia; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Mixed Dementias; AIDS Dementia Complex; Pick Disease of the Brain; Dementia, Multi-Infarct

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Building Better Caregivers Workshop Group (Experimental): Building Better Caregivers Workshop is a 6-week online self-management and skills building workshop. Participants receive the online workshop as soon as possible after randomization.
  Interventions: Behavioral: Building Better Caregivers Workshop
- Attention Control Group (Active Comparator): Participants will be offered the online workshop after the 12 month trial is completed if they so desire.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Building Better Caregivers Workshop — Workshops consist of small group or about 20-25 persons. Two peer co-facilitators (caregiver themselves) will guide workshop activities. Participants will receive a workshop booklet. Each week, participants will log on at least 2-3 times for a total time of approximately two hours. Participants do not require "real time" attendance at pre-determined times.
  Arms: Building Better Caregivers Workshop Group
Behavioral: Attention Control — Participants will receive two brief 15-30 minutes phone calls by study staff, and will receive a handbook on dementia and caregiver resources while they wait for the workshop.
  Arms: Attention Control Group

SUMMARY:
Rural caregivers face challenges of geographic isolation and lower health care access and quality. Many rural dementia caregivers experience serious health consequences due to caregiving responsibilities that can limit their ability to maintain their caregiving role. Thus, there is a pressing need for effective, scalable, and accessible programs to support rural dementia caregivers.

Online programs offer a convenient and readily translatable option for program delivery because they can be accessed by caregivers in the home and at the convenience of the user. Building Better Caregivers is an online 6-week, interactive, small-group self-management, social support, and skills-building workshop developed for caregivers of individuals with Alzheimer's disease or related dementia.

The investigators will conduct a hybrid effectiveness-implementation randomized controlled trial that will enroll and randomize 640 rural dementia caregivers into two groups: the intervention (workshop) group and the attention control group. Caregivers will be recruited throughout the United States. Primary outcomes will be caregiver stress and depressive symptoms. The investigators hypothesize that stress scores and depressive symptoms will be significantly improved at 12 months in the intervention group versus control group. The investigators will also identify key strengths (facilitators) and weaknesses (barriers) of workshop implementation. The investigators will use the RE-AIM implementation framework and a mixed methods approach to identify implementation characteristics pertinent to both caregivers and rural community organizations.

If the Building Better Caregivers workshop is proven to be effective, this research has the potential to open new research horizons, particularly on how to reach and effectively support isolated dementia caregivers in rural areas with an intervention that is scalable, even in low-resourced settings. If the workshop can achieve its goals with rural dementia caregivers, some of those most isolated, it would also be expected to be scalable in other low-resourced settings (e.g., in urban or suburban environments).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Caring for person with dementia
* Able to read and write in English
* Able to access the internet
* Providing care for ≥ 10 hours per week
* Reporting a minimum stress level of 4 or more on a 10-point scale
* Living in rural area of United States (self-identify or zip code is a Rural Urban Commuting Area Codes (RUCA) defined rural area)

Exclusion Criteria:

* Have an anticipated inability to complete the 12-month follow-up (e.g., planned travel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Yank, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The data to be shared will be individual participant data that underlie the results reported in published article(s), after deidentification (e.g., text, tables, figures, and appendices). The additional and related documents that will be available are study protocol and data dictionary. The data will become available beginning within 3 months of article publication and ending 5 years following article publication.The access criteria for the data to be shared will include researchers who provide a methodologically sound proposal in order to achieve aims in the approved proposal including performance of meta-analysis of individual participant data. Proposals should be directed to veronica.yank@ucsf.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years at a third party website (Link to be included later).
Supporting Information: Study Protocol
Time Frame: The data will become available beginning within 3 months of article publication and ending 5 years following article publication.
Access Criteria: The access criteria for the data to be shared will include researchers who provide a methodologically sound proposal in order to achieve aims in the approved proposal including performance of meta-analysis of individual participant data. Proposals should be directed to veronica.yank@ucsf.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years at a third party website (Link to be included later).

REFERENCES:
- [Derived] Santoyo-Olsson J, Covinsky KE, Cheng J, Gallagher Thompson D, Yank V. Utilization of home- and community-based services among rural family caregivers of persons with dementia: the role of the area deprivation index. Front Public Health. 2025 Oct 14;13:1688161. doi: 10.3389/fpubh.2025.1688161. eCollection 2025. PMID 41164840
- [Derived] Santoyo-Olsson J, Covinsky KE, Chesla CA, Lorig K, Gallagher-Thompson D, Cheng J, Luzanilla M, Macias Romo E, Aguayo Ramirez G, Karliner L, Yank V. Predictors of Psychological Distress Among Rural Family/Friend Caregivers of People Living With Dementia in the United States: Consequences of the COVID-19 Pandemic. J Gerontol B Psychol Sci Soc Sci. 2024 Feb 1;79(2):gbad164. doi: 10.1093/geronb/gbad164. PMID 37897201
- [Derived] Santoyo-Olsson J, Lorig K, Romo EM, Luzanilla M, Ramirez GA, Cheng J, Chesla C, Covinsky KE, Karliner L, Thompson DG, Fahrenwald N, Yank V. Study protocol for a hybrid effectiveness-implementation trial of the Building Better Caregivers online workshop for rural family/friend caregivers of people living with dementia. Contemp Clin Trials. 2022 Oct;121:106903. doi: 10.1016/j.cct.2022.106903. Epub 2022 Aug 31. PMID 36057375

RESULTS

PARTICIPANT FLOW:
Groups:
- Building Better Caregivers Workshop Group: The Building Better Caregivers Workshop is a 6-week online small group workshop. Participants received self-management and caregiving skills-building training and social support. They also received a workbook to keep.
- Attention Control Group: Attention control group participants received two 15-30 minutes phone calls and a handbook on dementia and caregiver resources.
Period: Overall Study
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Started | 304 | 114
Group Delivery Begins = Modified Intention to Treat Population | 300 | 109
1.5 Month Follow-up | 266 | 103
6-month Follow-up | 261 | 99
Completed | 196 | 69
Not Completed | 108 | 45
Not completed — Administratively removed prior to group delivery: unable to verify identify, duplicate, PLWD death | 4 | 5
Not completed — Planned study completion at 6-months. 2 final cohorts initiated with known follow up of 6 months. | 68 | 29
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Lost to Follow-up | 27 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group | Total
Number analyzed (Participants) | 304 | 114 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants in each group did not answer the age question.
  years
    number analyzed (Participants) | 302 | 112 | 414
    (all) | 61.79 (11.47) | 63.53 (10.57) | 62.26 (11.24)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 258 | 94 | 352
  Sex: Male | 42 | 20 | 62
  Sex: Prefers not to identify | 4 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-identified race and ethnicity.
  Participants
    White | 263 | 96 | 359
    Black/African American | 14 | 4 | 18
    Hispanic/Latino | 11 | 6 | 17
    American Indian/Native American/Alaska Native | 4 | 4 | 8
    Asian/Asian American | 0 | 1 | 1
    Native Hawaiian/Other Pacific Islander | 1 | 0 | 1
    More than one race | 3 | 0 | 3
    Other | 3 | 1 | 4
    Unknown or not reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 304 | 114 | 418
PHQ-8 [Mean (Standard Deviation); unit: units on a scale] — Depressive symptoms were measured using the 8-item Patient Health Questionnaire (PHQ-8), with score range 0-24 (higher score indicates worse depressive symptoms). Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 5.3 (4.4) | 5.9 (4.7) | 5.5 (4.5)
Stress [Mean (Standard Deviation); unit: units on a scale] — Stress was measured using the single-item visual numeric stress scale, with score range 0-10 (higher score indicates worse stress). Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 6.5 (1.8) | 6.8 (1.8) | 6.6 (1.8)
Caregiver Self-Efficacy [Mean (Standard Deviation); unit: units on a scale] — Caregiving self-efficacy was measured with the Caregiver Self-Efficacy scale (8 items), with score range, 1-10 (higher score indicates greater self-efficacy). The scale was not administered at follow-up assessments if caregivers reported that they were not providing caregiving at that time. Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 5.2 (1.8) | 5.1 (1.8) | 5.2 (1.8)
Zarit Care Burden [Mean (Standard Deviation); unit: units on a scale] — Care burden was measured with the Zarit Burden Interview (12 items), with score range, 0-24 (higher score indicates greater burden). The scale was not administered at follow-up assessments if caregivers reported that they were not providing caregiving at that time. Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 22.9 (8.6) | 22.6 (7.7) | 22.8 (8.3)
Self-Rated General Health [Mean (Standard Deviation); unit: units on a scale] — Poor self-rated health was measured using the single item Short Form Survey (SF-1) scale, with score range, 1-5 (higher score indicates worse health). Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 2.5 (0.9) | 2.6 (0.8) | 2.5 (0.9)
Loneliness [Mean (Standard Deviation); unit: units on a scale] — Loneliness was measured with the UCLA loneliness scale (3 items), with score range, 3-9 (higher score indicates greater loneliness). Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 6.0 (2.0) | 6.0 (1.9) | 6.0 (2.0)
Social Isolation [Mean (Standard Deviation); unit: units on a scale] — Social network was measured with the Lubben social network scale (6 items), with score range, 0-30 (higher score indicates greater network). Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 13.5 (5.6) | 13.4 (5.7) | 13.5 (5.6)
Healthcare Utilization [Mean (Standard Deviation); unit: days] — Healthcare utilization days was measured as emergency room and hospitalization days of use in the prior six months as a count, with range 0-180 days (higher count indicates more days). Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  days
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 0.23 (0.9) | 0.46 (1.9) | 0.3 (1.2)
Person with Dementia General Health (caregiver reported) [Mean (Standard Deviation); unit: units on a scale] — Poor self-rated health was measured using the single item Short Form Survey (SF-1) scale, with score range, 1-5 (higher score indicates worse health). Population: Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.
  units on a scale
    number analyzed (Participants) | 300 | 109 | 409
    (all) | 3.7 (1.0) | 3.7 (1.1) | 3.7 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Personal Health Questionnaire Depression (PHQ-8) Scale Score
Description: Personal Health Questionnaire Depression (PHQ-8) scale. The scale score is calculated by summing each item to produce a total score between 0 and 24, with higher scores indicating worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
units on a scale | 5.6 (4.1) | 5.8 (4.4)

2. Primary Outcome: Visual Numeric Stress Scale
Description: A visual numeric stress scale. The scale score ranges from 0 to 10, with higher score indicating worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
score on a scale | 5.9 (2.2) | 6.0 (2.1)

3. Secondary Outcome: Personal Health Questionnaire Depression (PHQ-8) Scale Score
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 261 | 99
units on a scale | 5.7 (4.6) | 7.1 (5.4)

4. Secondary Outcome: Visual Numeric Stress Scale Score
Description: A visual numeric stress scale. The scale score ranges from 0 to 10, with higher score indicating worse outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 261 | 99
units on a scale | 6.0 (2.2) | 5.9 (2.2)

5. Secondary Outcome: Short Caregiver Self-Efficacy Scale Score
Description: Short Caregiver Self-Efficacy scale (8-items). The scale scores is calculated by taking the mean of the items to produce a total score between 1 and 10, with higher scores indicating better outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
units on a scale | 5.4 (2.0) | 5.1 (1.6)

6. Secondary Outcome: Zarit Burden Interview-12 (ZBI-12) Scale Score
Description: Short form of the Zarit Burden Interview-12 (ZBI-12) scale (12-items). The scale score is calculated by summing each item to produce a total score between 0 and 24, with higher scores indicating worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
units on a scale | 21.9 (9.0) | 23.4 (7.3)

7. Secondary Outcome: Caregiver Self-rated General Health Score
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure SF-1 self-rated general health single item. The scale score ranges from 1 to 5, with higher scores indicating worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
units on a scale | 2.6 (0.9) | 2.7 (0.9)

8. Secondary Outcome: UCLA Loneliness Scale Score
Description: UCLA loneliness scale (3-items). The scale score is calculated by summing each item to produce a total score between 3 and 9, with higher scores indicating worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
units on a scale | 5.9 (2.0) | 5.4 (1.9)

9. Secondary Outcome: Lubben Social Isolation Scale Score
Description: Lubben Social isolation scale (6-items). The scale score is calculated by summing each item to produce a total score between 0 and 30, with lower scores indicating worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
units on a scale | 13.1 (5.7) | 13.8 (5.1)

10. Secondary Outcome: Caregiver Health Care Utilization
Description: 3-items measuring days of overnight hospitalizations, nursing home or other long-term care facility use, and hospital emergency room visits from the Health and Retirement Study, modified time frame from self-report for past 12 months to self-report for past 6 months; scored as single items; with higher scores indicating worse outcome. Scores range from 0-180.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
days | 0.30 (1.3) | 0.84 (3.1)

11. Secondary Outcome: Person With Dementia General Health Score as Reported by Caregiver
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) measure SF-1 caregiver-reported general health single item. The scale score ranges from 1 to 5, with higher scores indicating worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
Number analyzed (Participants) | 196 | 69
units on a scale | 3.8 (1.0) | 3.8 (1.0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Building Better Caregivers Workshop Group | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/304 | 1/114
Serious Adverse Events (participants affected / at risk) | 0/304 | 1/114
Other Adverse Events (participants affected / at risk) | 0/304 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Building Better Caregivers Workshop Group (N=304) | Attention Control Group (N=114)
natural disaster (General disorders) | 0 | 1 — One death unrelated to the study occurred (i.e., an "act of God" event). During a state of emergency caused by massive rainstorms and flooding, a tree fell onto the roof of the participant's house and crushed her when she was in bed asleep.

LIMITATIONS AND CAVEATS:
Randomization occurred 2 weeks before group delivery to allow for mailing of books and scheduling calls. During this run-in period 9 participants were administratively dropped: 4 in intervention group, due to death of person with dementia (2), being a duplicate (1), and inability to verify identity (1); 5 in control group, due to death of their person (3), death of caregiver in natural disaster (1), and being paid caregiver (1). Thus, the modified ITT analysis included 409 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Protocol and SAP (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT04428112/Prot_SAP_000.pdf
  • Study Protocol: Revised protocol (randomization plan subsection) (2019-08-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT04428112/Prot_001.pdf
  • Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT04428112/ICF_002.pdf